CLINICAL TRIAL: NCT01660919
Title: Vascular and Metabolic Effects of Rosuvastatin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Kwang Kon Koh, professor, Gachon University Gil Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GMC-201105
Record Dates: First submitted 2012-08-08; First posted 2012-08-09 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2012-08

CONDITIONS: Hypercholesterolemia
Keywords: insulin resistance
MeSH Terms: conditions — Hypercholesterolemia; Insulin Resistance | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- placebo (Placebo Comparator): placebo
  Interventions: Drug: placebo
- rosuvastatin 5 (Active Comparator): rosuvastatin 5 mg
  Interventions: Drug: rosuvastatin
- rosuvastatin 10 (Active Comparator): rosuvastatin 10 mg
  Interventions: Drug: rosuvastatin
- rosuvastatin 20 (Active Comparator): rosuvastatin 20 mg
  Interventions: Drug: rosuvastatin

INTERVENTIONS:
Drug: placebo
  Arms: placebo
Drug: rosuvastatin
  Arms: rosuvastatin 10; rosuvastatin 20; rosuvastatin 5

SUMMARY:
The investigators hypothesize that rosuvastatin does-dependently worsens insulin sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* hypercholesterolemia

Exclusion Criteria:

* overt liver disease, chronic renal failure, hypothyroidism, myopathy, uncontrolled diabetes (HbA1c > 9%), severe hypertension, stroke, acute coronary events, coronary revascularization within the preceding 3 months, or alcohol abuse

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2011-10; Primary Completion 2013-01 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
flow-mediated dilation | 8 weeks of treatment

SECONDARY OUTCOMES:
insulin resistance | 8 weeks of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Gil Medical Center, Incheon, South Korea